CLINICAL TRIAL: NCT05018702
Title: A Prospective, Single-arm, Single-center Phase II Clinical Study of Recombinant Humanized Anti-HER2 Monoclonal Antibody-AS269 Conjugate (ARX788) in the Treatment of HER2-positive Breast Cancer Patients With Brain Metastases
Brief Title: ARX788 in HER2-positive Breast Cancer Patients With Brain Metastases
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xichun Hu, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACE-Breast-06
Record Dates: First submitted 2021-08-22; First posted 2021-08-24 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: HER2-positive, Metastatic Breast Cancer
Keywords: ARX788; HER2-positive breast cancer; Brain metastasis
MeSH Terms: conditions — Breast Neoplasms; Brain Neoplasms | interventions — ARX788

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ARX788 (Experimental)
  Interventions: Drug: ARX788

INTERVENTIONS:
Drug: ARX788 — 1.5 mg/kg IV infusion on Day 1 of each 21-day treatment cycle.

SUMMARY:
A Phase 2 Study of ARX788 in HER2-positive, Metastatic Breast Cancer Patients whose Disease is resistant or refractory to Tyrosine kinase inhibitors (TKI).

DETAILED DESCRIPTION:
This is an open-label, single arm, phase 2 study of ARX788 in HER2-positive, metastatic breast cancer patients whose disease is resistant or refractory to TKI. The ARX788 will be administered every 3 weeks (Q3W) intravenous (IV) infusion. In this study, Simon's two-stage design is used. Subjects received treatment until disease progression, intolerable toxicity, withdrawal from the study, or discontinuation judged by the investigator. Drug efficacy and safety data will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years, and ≤75 years, male or female;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0~2;
* Breast cancer patients diagnosed as HR arbitrary/HER2-positive by pathological examination;
* Metastatic breast cancer subjects previously treated with trastuzumab, taxane and EGFR-TKI-containing regimens;
* MRI confirmed brain metastasis with at least one intracranial parenchymal untreated metastatic lesion;
* Mannitol, bevacizumab, or hormone therapy is allowed before enrollment;
* Adequate organ functions;
* Acute toxicities from any prior therapy, surgery, or radiotherapy must have resolved to Grade ≤1.
* Patients who participate in the trial voluntarily, sign an informed consent, have good compliance and are willing to comply with the follow-up visit.

Exclusion Criteria:

* Pneumomeningeal metastases or cystic metastases confirmed by MRI or lumbar puncture;
* Uncontrolled third space effusion;
* Previous treatment with T-DM1 or other HER2-ADC drugs;
* Received a whole-brain radiotherapy, chemotherapy, or surgery within 2 weeks prior to the first dose of ARX788, or trastuzumab-targeted therapy or endocrine therapy within 1 week, or palliative radiotherapy for bone metastases within 2 weeks;
* Prior history of interstitial pulmonary disease requiring hormone therapy, drug-induced interstitial pulmonary disease, radiation pneumonia, or current clinically active interstitial pulmonary disease;
* Suffering from keratitis, corneal diseases, retinal diseases or active eye infections that require intervention;
* Unwilling or unable to stop wearing contact lenses for the duration of the study;
* Participated in other clinical trials within 2 weeks prior to enrollment;
* Receiving any antitumor therapy for any other tumor, bevacizumab for the control of brain edema and bisphosphonates for the treatment of bone metastases or the prevention of osteoporosis are the exception;
* With a history of any malignancies other than breast cancer in the past 5 years, excluding cured cervical carcinoma in situ, basal cell carcinoma of the skin or squamous cell carcinoma of the skin;
* Cardiac insufficiency;
* Uncontrolled hypertension;
* History of allergic reactions to any component of ARX788, or with a history of protein drug allergy, a history of specific allergies (asthma, rheumatism, eczematous dermatitis), or a history of other severe allergic reactions, who are unsuitable for ARX788 treatment as per the investigator's judgments;
* Pregnancy or lactation;
* History of immunodeficiency, including HIV-positive, or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation;
* Current known active infection with human immunodeficiency virus (HIV), hepatitis B virus, hepatitis C virus or syphilis;
* History of neurological or psychiatric disorder, including epilepsy or dementia;
* Suffering severe or uncontrolled systemic diseases.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2021-07-14 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Central nervous system (CNS) clinical benefit rate (CBR) | 2 years
  CNS CBR is defined as the percentage of subjects who have achieved complete response, partial response, and stable disease according to the Response Assessment in Neuro-Oncology Brain Metastases (RANO-BM) criteria

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 2 years
  PFS is defined as the time between date of first dose of study therapy and date of progression or death, whichever occurs first, will be computed for response evaluable subjects. Subjects will be censored at time of subsequent therapy
Overall survival (OS) | 2 years
  Overall survival (OS) is defined as the time from first dose of study therapy to the date of death (any cause). Subjects who are alive will be censored at the last known time that the subject was alive
Site of first progression | 2 years
  Record the organs where the disease first progressed during the study
The number of subjects experiencing adverse events | 2 years
  Patient safety and adverse events (AEs) will be evaluated using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v.5.0. All AEs and serious adverse events (SAEs) will be assessed to determine the safety and tolerability of the treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li T, Lin M, Wang B, Zhao M, Cao J, Wang L, Tao Z, Jin J, Miao H, Gong C, Zhao Y, Peng W, Hu X, Zhang J. Efficacy and safety of ARX788 for individuals with HER2-positive breast cancer and brain metastases (ACE-Breast-06): a single-arm, phase 2 trial in China. EClinicalMedicine. 2025 Oct 30;90:103614. doi: 10.1016/j.eclinm.2025.103614. eCollection 2025 Dec. PMID 41245540